CLINICAL TRIAL: NCT02811120
Title: An Observational Follow up Study of a Phase II/III, Open Label, Randomised Study of the Safety, Reactogenicity and Immunogenicity of a Single Dose of Meningococcal ACWY Conjugate Vaccine (Menveo, Glaxosmithkline or Nimenrix, Pfizer) in Adolescents Who Were Primed With Meningitec, Menjugate or Neisvac-C During Preschool Vaccination
Brief Title: PRIME Follow up - Quadri Meningo Vacinees
Acronym: PRIMEfollowup
Status: Completed | Type: Observational
Sponsor: Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: PRIMEfollowup
Record Dates: First submitted 2016-06-15; First posted 2016-06-23 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2018-08

CONDITIONS: Meningococcal Disease
Keywords: meningococcal; conjugate; vaccine; quadrivalent; meningococcal quadrivalent conjugate vaccine
MeSH Terms: conditions — Meningococcal Infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — serology samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- single arm: single venepuncture
  Interventions: Other: venepuncture only

INTERVENTIONS:
Other: venepuncture only — single venepuncture

SUMMARY:
A previous cohort of 93 clinical trial participants received quadrivalent meningococcal conjugate vaccine, which includes strains ACW and Y, in their teenage years. The vaccine also contains components of diphtheria and tetanus which are linked to the meningitis components, in a process called conjugation, to improve their effectiveness.

Participants are now aged 19-25 and will be invited to take part in this study, which will assess antibody persistence over time. This will provide information about the duration of protection by relating current antibody levels to those measured in the previous study, and will underpin the national immunisation schedule in providing optimal immunisation schedule. As well as the meningitis antibodies the investigators will assess diphtheria and tetanus antibody levels.

The study will involve a single blood test of up to 8mL. Participants will be informed of their results and any with an antibody level that does not infer protection against strain W will be offered an extra dose of vaccine as part of a duty of care.

The study will involve a single blood test of up to 8mL. Participants will be informed of their results and any with an antibody level that does not infer protection against strain W will be offered an extra dose of vaccine.

DETAILED DESCRIPTION:
The UK was the first country in the world to introduce the meningococcal serogroup C conjugate vaccine (MCC) into its routine immunisation schedule in 1999. This very effectively reduced the incidence of disease, which was highest in those younger than 1 year through its routine use in the infant immunisation schedule, and those aged around 15-17 years through a catch up campaign . Subsequently, the meningococcal vaccination schedule has undergone several revisions, including:

* 2006 - a reduction in the number of doses given to infants from the manufacturer advised three to the JCVI instructed two with the combination of the MCC dose in the second year of life with the Hib vaccine, in the form of Menitorix
* 2013 - a further reduction to a single dose in infancy and the introduction of a booster in teenage years due to studies demonstrating that antibody persistence was short lived through childhood
* 2015 - the amendment of the teenage booster dose from MCC to a quadrivalent meningococcal conjugate vaccine to address the increasing incidence of serogroup W disease in this age group (PHE website - Meningococcal data), and the introduction of Bexsero into the infant schedule ostensibly to address meningococcal B disease but with the potential for cross protection against other serogroups, which is currently being assessed in another NVEC study.
* 2016 - removal of the MCC at 3 months of age.

Given the previous demonstration of poor antibody persistence of MenC antibodies two years following the 2006 schedule, with only 43%, 22% and 23% of children achieving SBA titres ≥8 two years following a booster dose of Menitorix™ when primed with NeisVac-C™, Menjugate™ and Meningitec™, respectively, there is concern about the protection afforded by the quadrivalent vaccine administered at around 14 years of age, and whether this will provide protection into young adulthood when the risk of disease is high.

In a previous study by this group (Eudract number 2010-022505-18) , adolescents aged 16-19 years were randomised to receive one of two licensed meningococcal ACWY conjugate vaccines:

1. Menveo™ (GSK) This vaccine contains bacterial capsular oligosaccharides for serogroups A, C, W, and Y conjugated to a protein carrier, CRM197, which is a nontoxigenic natural variant of diphtheria toxin. The MenACWY vaccine has been tested in several age groups and has been shown to be generally well tolerated and immunogenic. Menveo™ is indicated for use in those from 2 years of age and in those at risk.
2. Nimenrix (Pfizer) This vaccine contains bacterial capsular oligosaccharides for serogroups A, C, W, and Y conjugated to Tetanus Toxoid (TT). This MenACWY-TT vaccine has been tested in several age groups and has been shown to be safe and immunogenic. It is indicated for use from 12 months of age and in those at risk.

The cohort included in this study was one of the first to receive meningococcal C conjugate vaccine as young children, and subsequently to have the booster in the form of meningococcal quadrivalent (ACWY) conjugate vaccination at age 16-19 years. This group of 93 young adults, now aged 20-24 years, provides a unique opportunity to study the persistence of meningococcal serogroup-specific antibodies over time. This is particularly important given the recent increases in incidence of meningococcal W disease which prompted the amendment of the national schedule to include a booster of the meningococcal quadrivalent vaccine in teenage years.

ELIGIBILITY:
Inclusion Criteria:

* Individual is willing and able to give written informed consent for participation.
* Individual was originally enrolled in the randomised parallel group study of quadrivalent meningococcal vaccination.

Exclusion Criteria:

* Known bleeding diathesis (or any condition that may be associated with a prolonged bleeding time).
* Any other significant condition or circumstance which, in the opinion of the investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Health volunteers who previously took part in a clinical trial of meningococcal quadrivalent vaccine
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Serum bactericidal antibody (SBA) assays | single timepoint per participant, within the 12 month study timeframe
  Strains C11, F8238, M01 240070, M03 241125

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Coates, PhD, Study Chair — Public Health England

IPD SHARING:
Plan to Share IPD: No
No plan to share IPD